CLINICAL TRIAL: NCT03017807
Title: A PhaseⅠ,Open-label, Single-center Study to Evaluate Safety and Pharmacokinetics of Recombinant Anti-Epidermal Growth Factor Receptor (EGFr) Antibody in Patients With Metastatic Colorectal Cancer
Brief Title: Safety and Pharmacokinetics of Recombinant Anti-EGFr Antibody in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Kelun Pharmaceutical Co., Ltd (Industry)
Collaborators: 307 Hospital of PLA (Other)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL140-I-01-CTP
Record Dates: First submitted 2016-12-29; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recombinant Anti-EGFr Antibody (Experimental): Low-dose level patients received cetuximab initial dose 100 mg/m2 and 4 weeks later 250 mg/m2 weekly maintenance.High-dose level patients received cetuximab initial dose 400 mg/m2 and 4 weeks later loading 400 mg/m2 and 250 mg/m2 weekly maintenance.
  Interventions: Biological: Recombinant Anti-EGFr Antibody

INTERVENTIONS:
Biological: Recombinant Anti-EGFr Antibody — Low-dose level patients received cetuximab initial dose 100 mg/m2 and 4 weeks later 250 mg/m2 weekly maintenance to the disease progression or unacceptable toxicity or death or withdraw informed consent.High-dose level patients received cetuximab initial dose 400 mg/m2 and 4 weeks later loading 400 mg/m2 and 250 mg/m2 weekly maintenance to the disease progression or unacceptable toxicity or death or withdraw informed consent.

SUMMARY:
A single-central,open-label,safety,pharmacokinetics,phase I study. Biological:Recombinant Anti-EGFr Antibody Two dose levels: Low-dose level patients received initial dose 100 mg/m2 and 4 weeks later 250 mg/m2 weekly maintenance to the disease progression or unacceptable toxicity or death or withdraw informed consent.High-dose level patients received cetuximab initial dose 400 mg/m2 and 4 weeks later loading 400 mg/m2 and 250 mg/m2 weekly maintenance to the disease progression or unacceptable toxicity or death or withdraw informed consent.

DETAILED DESCRIPTION:
Two dose levels were tested: Recombinant Anti-EGFr Antibody Low-dose level patients received initial dose 100 mg/m2 and 4 weeks later 250 mg/m2 weekly maintenance to the disease progression or unacceptable toxicity or death or withdraw informed consent.High-dose level patients received cetuximab initial dose 400 mg/m2 and 4 weeks later loading 400 mg/m2 and 250 mg/m2 weekly maintenance to the disease progression or unacceptable toxicity or death or withdraw informed consent. Dose limiting toxicity (DLT) was defined as: grade 4 or 3-time grade 3 cutaneous toxicity,successive 3-time infusion suspension due to grade 3 cutaneous toxicity,any other ≥grade 3 adverse reaction or acute pneumonia, interstitial pneumonia, and other lung diseases.

Cohorts of 3 patients receive single dose of low-dose group of Recombinant Anti-EGFr Antibody. If the ratio of the dose limiting toxicity (DLT) after a single dose is not more than a third, then high-dose group can be treated.After high-dose(initial dose 400 mg/m2, iv., 2 h),safety will be observed and blood sampling will be taken for a single dose pharmacokinetic analysis.After 4-week continuous administration (loading dose 400 mg/m2, iv., 2 h; maintenance dose 250 mg/m2, iv, 1 h, q1w) until disease progression, unacceptable toxicity reaction, death or revocation of informed consent.As the blood concentration reach steady state, blood sampling will be collected for steady-state pharmacokinetic analysis, for 1 week.After completion of the steady-state pharmacokinetics,patients can receive chemotherapy,and safety (including immunogenicity) and curative effect will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Ages eligible for study between 18 Years and 75 Years.
2. Confirmed histological diagnosis of colorectal cancer.
3. Subjects with advanced/metastatic Colorectal Cancer(CRC) who have failed to the irinotecan- ,oxaliplatin- and fluoropyrimidine-based regimens or been intolerant to irinotecan or rejected the chemotherapy.
4. Eastern Cooperative Oncology Group (ECOG) of 0 or 1.
5. Subjects must have a life expectancy of at least 12 weeks.
6. Patients with at least one evaluable lesion (evaluable disease) by the RECIST criteria.
7. Adequate renal function (creatinine ≤ 1.5 x UNL), liver function (total bilirubin ≤ 1.5 x UNL, alanine aminotransferase(ALT)< 2.5 x UNL, aspartate aminotransferase(AST) < 2.5 x UNL or ≤ 5 x UNL if hepatic metastasis) and leucocytes ≥ 3×10^9, absolute neutrophil count ≥ 1.5×10^9/L, platelets > 80×10^9/L, haemoglobin ≥ 9 g/dl. Electrolyte: in the normal range, or abnormal but no clinical significance (judged by the researchers), allow to give supplements to correct the electrolyte.
8. Both women of child-bearing potential and sexually active men must agree to use adequate contraception prior to study entry and for the duration of study participation and for 90 days after the conclusion of study therapy.
9. Patients who have capable to understand the procedure and methods of the study,are willing to strictly follow the protocol and sign the the informed consent.

Exclusion Criteria:

1. Previous therapy with anti-EGFR drugs.
2. Patients who are receiving other accompanying antineoplastic therapy (including antitumor treatment with traditional Chinese medicine), long-term systemic immune therapy, or hormone therapy except for physiological replacement therapy (for example, people with thyroid hypofunction receive the thyroid hormone).
3. Radiotherapy or surgery (except always diagnostic biopsy).
4. Patients with known cerebral metastasis or leptomeningeal metastasis.
5. Any other malignant tumour in the last five years, except for suitably treated in situ cervical carcinoma or basal cell carcinoma.
6. Clinically significant cardiovascular disease, such as heart failure (NYHA Ⅲ-Ⅳ), uncontrolled coronary heart disease, cardiomyopathy, cardiac arrhythmias, hypertension (> 140/90 mmHg), myocardial infarction in the last half year, echocardiogram showed ejection fraction < 50%.
7. Patients with any symptom of acute or subacute bowel obstruction and/or inflammatory bowel disease.
8. Patients with known active and severe infections(> grade 2, National Cancer Institute Common Toxicity Criteria(NCI-CTC) adverse effect(AE) V. 4.03), including active tuberculosis(TB).
9. HIV infection or active hepatitis B or hepatitis C.
10. Uncontrolled diabetes (> grade 2, NCI-CTC AE V. 4.03), severe lung disease (acute lung disease, pulmonary fibrosis that affect the lung function, and interstitial lung disease), liver failure.
11. Patients with blood coagulation dysfunction as following situation: prothrombin time (PT) ≥ 1.5 x UNL, thrombin time (TT) ≥ 1.5 x UNL, the part activated clotting time (APTT) ≥ 1.5 x UNL.
12. Patients who have blood transfusion, or use the g-csf cytokines etc in the last 10 days.
13. Known hypersensitivity to any component of pretreated product.
14. Pregnancy or breastfeeding.
15. Patients with known drug and/or alcohol abuse.
16. Patients with a clear history of neurological or psychiatric disorders, including epilepsy or dementia.
17. Patient participation in another clinical trial or receive other research drugs during the previous 4 weeks.
18. Patients with a medical or mental abnormalities unable to give informed consent.
19. Lack of legal behavior ability or limited legal behavior ability.
20. Other factors that may affect the efficacy or safety evaluation of this study assessed by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity. | 4 weeks after the single dose
  Dose limiting toxicity (DLT) was defined as: grade 4 or 3-time grade 3 cutaneous toxicity,successive 3-time infusion suspension due to grade 3 cutaneous toxicity,any other ≥grade 3 adverse reaction or acute pneumonia, interstitial pneumonia, and other lung diseases.

SECONDARY OUTCOMES:
Change from baseline in serum antibody and its neutralizing ability | Prior to the single dose on day 1 and on the 1st day of 1、2、4、6、9 week after the first administration until 1 month after the last administration.
Pharmacokinetics (PK): Area Under the Concentration Curve (AUC) of anti-EGFR antibody after single dose and under the stable blood concentration. | 4 weeks after the single dose and 1 week under the stable blood concentration after weekly administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Kelun Pharmaceutical Co., Ltd., Chengdu, China

IPD SHARING:
Plan to Share IPD: No